CLINICAL TRIAL: NCT02114580
Title: Brain Plasticity Following Aerobic Exercise in Patient With Mild Cognitive Impairment: Neuroimaging Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0051-14-TLV
Record Dates: First submitted 2014-03-31; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-03

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; exercise; brain plasticity; FMRI
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise (Experimental)
  Interventions: Other: physical training
- stretching exercise (Active Comparator)
  Interventions: Other: physical training

INTERVENTIONS:
Other: physical training — Participants in both the aerobic and stretching groups will carry out their activity routines 3 d/wk for 45 to 60 minutes per session for 4 months. Training will be on "one on one" basis, where each participant will be supervised by an experienced trainer at the participant's home.Aerobic intervention protocol: subjects will practice with stationary bicycle. Exercise intensity will be monitored through wireless HR monitor. Participants will be also monitored for the intensity of their workouts by the Borg's Rating of Perceived Exertion and the "talk" test (a subjective method for estimating of appropriate cardiorespiratory exercise intensity).
  Stretching exercise protocol: Participants in the stretching control group will carry out a prescribed routine of stretching and balance exercises.

SUMMARY:
The proposed study aims to explore brain mechanisms mediating the cognitive benefits of aerobic exercise in patients with mild cognitive impairment- a prodromal stage of Alzheimer disease. We will perform FMRI experiments, as well as laboratory and behavioral tests that will advance our knowledge about the nature of these mechanisms. Participants will participate in individual- tailored aerobic training program. Pre and post evaluation will identify brain changes following the training using advanced techniques of brain imaging. Cognitive performance will be assessed prior and at the end of the program, as well as endocrine markers reflecting improvement in learning abilities. Moreover, demonstrating cortical plasticity in subjects with aMCI has tremendous practical significance for these subjects .

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI), a prodromal stage of Alzheimer disease (AD), refers to a transitional state between the cognition of normal aging and dementia such AD. To date, therapeutic approaches to AD are symptomatic and of modest efficacy. Nontheless, recent studies in animal models or healthy subjects, have shown that aerobic exercise affect brain plasticity. The current proposal aims at exploring the brain mechanisms mediating the cognitive benefits of aerobic exercise in patients with amnestic MCI (aMCI),in compare to a control group of subjects with aMCI receiving stretching exercise. More specifically, we aim to perform two fMRI experiments, that will advance our knowledge about the nature of mechanism of the cognitive benefit resulting of aerobic exercise. Our preleminary results suggest that subjects with aMCI show different hierarchy of reliable responses when processing long time scales in auditory task. Therefore, in the first experiment, we will evaluate how these patterns of temporal hierarchy of language processing are affected by aerobic exercise. Next, we will explore whether aerobic exercise affect memory enocoding task, which rely on areas in the medial temporal lobe who bear a heavy neuropathological burden in MCI. The insights gained from the study may have important clinical implications for patients who are at the early stages of Alzheimer's disease

ELIGIBILITY:
Inclusion Criteria:

* Only patients at the age of 60-90 who have met criteria for a diagnosis of MCI will be included.
* Participants will be both men and women, and this factor is not specifically addressed.

Exclusion Criteria:

* Patients with any significant medical (i.e. cardiac), neurological (other than MCI) illness will be excluded from the study.
* Medical and neurological illnesses will be ruled out by physical and neurological examinations, reports of the patients' treating physicians and medical records.
* The experiments will be undertaken in compliance with the safety guidelines for MRI research. Based on initial fMRI screening questionnaires, subjects will be excluded if they indicate any risk factor on these questionnaires.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
functional Magnetic Resonance Imaging | two weeks prior to intervention

SECONDARY OUTCOMES:
Neuropsychological assessment | two weeks prior to intervention

OTHER OUTCOMES:
Cardiorespiratory fitness assessment, Serum concentration of BDNF | two weeks prior to intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Lerner, PhD, Principal Investigator — Functional Brain Center, Wohl Institute for Advanced Imaging, Tel-Aviv Sourasky Medical Center, Tel-Aviv, Israel
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel